CLINICAL TRIAL: NCT06406569
Title: Home RehabGym: a Qualitative and Usability Evaluation of Advanced Technologies for Home Upper Limb Neurorehabilitation Post-stroke
Brief Title: A Qualitative and Usability Evaluation of Advanced Technologies for Home Upper Limb Neurorehabilitation Post-stroke
Acronym: Home RehabGym
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tan Tock Seng Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DSRB 2023/00527
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Stroke
Keywords: Technology-aided; Upper limb rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: The study design is a pilot, clinical feasibility, assessor-blinded trial to evaluate the feasibility of Home RehabGym concept through deployment of three rehabilitation devices at patients' homes: MyoPanda, H-Man and ReHandyBot.
  During the 6 weeks training at home phase, patients will be provided with two devices at any one time: with only the MyoPanda being used by the patient for 6 weeks. The H-Man and ReHandyBot will stay with the patient for 3 weeks (i.e. 21 days) each and then alternate.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Home Robotics Upper Limb Training (Other): The patients will first familiarize in the clinic with the 3 devices (H-MAN, ReHandyBot and MyoPanda) with initial assistance of the therapists and then take the devices home for independent, self-administered training under caregiver supervision.
  During the 6 weeks training (home phase), patients will be provided with two devices at any one time: with only the MyoPanda being used by the patient for 6 weeks. The H-MAN and ReHandyBot will stay with the patient for 3 weeks (i.e., 21 days) each.
  Interventions: Device: H-Man Robot; Device: ReHandyBot; Device: MyoPanda

INTERVENTIONS:
Device: H-Man Robot — The HMAN is certified as a CE class 2A upper limb rehabilitation robot suitable for hospital, clinic and home-based use in 2020 by Health Sciences Authority, Singapore. It has since been employed in post-stroke neurorehabilitation therapy and assessment of sensorimotor functions in stroke patients.
Device: ReHandyBot — ReHandyBot is the portable version of ReHapticKnob a robot developed at ETH Zurich that provides neurocognitive therapy, focusing on hand opening and closing movements as well as prono-supination of the forearm.
Device: MyoPanda — MyoPanda is a passive wrist/hand device which patients use to train the hand and wrist function by controlling a virtual avatar with EMG activity measures.

SUMMARY:
Due to limited resources such as the low therapist to patient ratio or high costs associated to rehabilitation therapy, providing higher therapy dose to patients after discharge is highly challenging. This often results in non-use of the impaired limb as a result of the decreased therapy dose, causing partial loss of the functional improvements previously gained during early rehabilitation.

In this study, the investigators plan to pilot the HomeRehab Gym concept via the deployment of three rehabilitation devices at patients' homes: MyoPanda, H-Man and ReHandyBot.

DETAILED DESCRIPTION:
Previous research has proven that technology-aided upper limb rehabilitation is non-inferior in terms of feasibility and efficacy when compared to conventional therapy in stroke patients. These rehabilitation devices can be set up as a 'rehabilitation gym' (RehabGym), where patients can interact with several devices that target different body and rehabilitation domains and, thus allows for a holistic and complementary therapy.

Despite recent studies having shown that training with a RehabGym under reduced supervision in a hospital is not only feasible but also equally beneficial in terms of clinical outcomes, however, a RehabGym has never been set up at a patient's home to the best of our knowledge.

This study aims to investigate the feasibility and safety of a RehabGym at home concept using three different upper-limb technologies (H-Man, ReHandyBot, MyoPanda) that are established, clinically tested and allow for on-demand therapy. Objective measures of clinical efficacy will also be examined, and cost-analysis to determine the economic feasibility of a commercial implementation of RehabGym at home in the future will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical stroke (ischaemic or haemorrhagic) confirmed by admitting doctors and CT, CT angiography or MRI brain imaging
2. Age 21 to 80 years, both males and females
3. At least 28 days post-stroke
4. Upper limb motor impairment of Fugl-Meyer Assessment (FMA) scale 20 to 50
5. Montreal Cognitive Assessment (MoCA) > 21/30
6. Ability to sit supported and continuously for 60 minutes
7. Stable home abode with enough space to place technologies
8. Has a carer/next of kin to supervise home-based exercises

Exclusion Criteria:

1. Functional impairment of the upper limb due to other pathologies
2. Medical conditions incompatible with research participation: uncontrolled medical illnesses (hypertension or diabetes, ischaemic heart disease, congestive heart failure, bronchial asthma, severe /untreated depression, agitation, end stage renal/liver/heart/lung failure, unresolved cancers)
3. Anticipated life expectancy of less than 6 months
4. Pacemakers and other active implants
5. Active seizures within 3 months
6. Local factors potentially worsened by intensive technology-aided upper-limb therapy and computer-based training:

   * Spasticity - modified Ashworth Scale MAS > 2 of any upper limb muscle groups
   * Severe pain in affected arm - Visual Analogue Scale for pain VAS > 5/10
   * Skin wounds
7. Cognitive impairment precluding study participation
8. Severe visual impairment or visual neglect affecting ability to use technologies
9. History of dementia, depression or behavioural problems
10. Pregnant or lactating females will not be allowed to participate

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07-31 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Compliance Rates | Through study's data collection period, up to 2 years.
  Using cloud data from vendor, time (min/hours) of robot (H-Man, ReHandyBot, MyoPanda) usage

SECONDARY OUTCOMES:
Fugl Meyer Motor Assessment (FMA) | Weeks 0 (baseline), 3 (mid-intervention assessment), 6 (post-intervention assessment), 12 (1st follow-up assessment), 24 (last follow-up assessment)
  Change in Fugl Meyer Motor Assessment score in the affected arm, minimum 0, maximum 66, with higher scores indicating better function
Action Research Arm Test (ARAT) | Weeks 0 (baseline), 3 (mid-intervention assessment), 6 (post-intervention assessment), 12 (1st follow-up assessment), 24 (last follow-up assessment)
  Functional and dexterity score for upper extremities, minimum 0, maximum 57; with higher score indicating better function
System Usability Scale (SUS) | Weeks 3 (mid-intervention assessment), 6 (post-intervention assessment))
  For evaluation of the different robots' (H-Man, ReHandyBot, MyoPanda) perceived usability, scaled from 1 (Strongly disagree) to 5 (Strongly Agree)
Hr-QOL scales using SS-QOL (Stroke specific Quality of Life scale) | Weeks 0 (baseline), 6 (post-intervention assessment), 12 (1st follow-up assessment), 24 (last follow-up assessment)
  Quality of life scale specific to stroke patients, minimum 49, maximum 245; with higher scores indicating better function.
Box and Block Test (BBT) | Weeks 0 (baseline), 3 (mid-intervention assessment), 6 (post-intervention assessment), 12 (1st follow-up assessment), 24 (last follow-up assessment)
  Measures unilateral gross manual dexterity.

CONTACTS AND LOCATIONS:
Overall Officials: Kuah Wee Keong Christopher, Principal Investigator — Tan Tock Seng Hospital
Locations (1):
- Tan Tock Seng Hospital, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No